CLINICAL TRIAL: NCT01966419
Title: Multicenter, Randomized Phase 2B Study to Evaluate the Efficacy, Safety and Tolerability of OCR-002 (Ornithine Phenylacetate) in Hospitalized Patients With Cirrhosis and Associated Hyperammonemia With an Episode of Hepatic Encephalopathy (STOP-HE Study)
Brief Title: Phase 2B Efficacy/Safety of Ornithine Phenylacetate in Hospitalized Cirrhotic Patients With Hepatic Encephalopathy (STOP-HE)
Acronym: STOP-HE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCR002-HE209; 2013-005412-10 (EudraCT Number)
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Acute Episode of Overt Hepatic Encephalopathy; Hepatic Encephalopathy
Keywords: hepatic encephalopathy; hyperammonemia; cirrhosis; ornithine phenylacetate; OCR-002
MeSH Terms: conditions — Hepatic Encephalopathy; Hyperammonemia; Fibrosis | interventions — ornithine phenylacetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: While the study was double-blind (participant and investigator blinded), the care provider and outcomes assessor were also blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ornithine phenylacetate (Active Comparator): Participants receive ornithine phenylacetate for up to 5 days via continuous IV infusion in addition to standard of care (SOC)
  Interventions: Drug: ornithine phenylacetate
- Placebo (Placebo Comparator): Participants receive matching placebo up to 5 days via continuous IV infusion in addition to SOC
  Interventions: Drug: placebo intravenous infusion

INTERVENTIONS:
Drug: ornithine phenylacetate — Ornithine phenylacetate for continuous IV infusion at dose levels predicated on level of hepatic decompensation
  Other Names: OCR-002
  Arms: Ornithine phenylacetate
Drug: placebo intravenous infusion — Placebo for continuous IV infusion that is visually identical to the experimental product
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether ornithine phenylacetate can speed recovery from an acute hepatic encephalopathy episode requiring hospitalization in cirrhotic patients.

DETAILED DESCRIPTION:
The primary objectives of the study were to evaluate the efficacy of OCR-002 for treatment of an acute hepatic encephalopathy (HE) episode in cirrhotic patients requiring hospitalization and the safety and tolerability of OCR-002 in hospitalized cirrhotic patients with an acute episode of HE.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with an acute episode of hepatic encephalopathy as complication of cirrhosis
* Elevated venous ammonia

Exclusion Criteria:

* Renal failure with serum creatinine > 3 mg/dL or need for dialysis
* Molecular Adsorbent Recirculation System utilized
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Chair — Ocera Therapeutics, Inc.
Locations (102):
- United States (32):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Coronado, California
  - Los Angeles, California
  - San Francisco, California
  - New Haven, Connecticut
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Glenview, Illinois
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Columbia, Missouri
  - Newark, New Jersey
  - Buffalo, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (6):
  - Kingswood, New South Wales
  - Adelaide, South Australia
  - Bedford Park, South Australia
  - Melbourne, Victoria
  - Melbourne
  - Parkville
- Austria (2):
  - Graz
  - Vienna
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Sofia, Bulgaria
- Czechia (3):
  - Brno
  - Prague
  - Ústí nad Labem
- Denmark (4):
  - Aarhus
  - Copenhagen
  - Esbjerg
  - Hvidovre
- Tartu, Estonia
- France (10):
  - Bordeaux
  - Grenoble
  - La Roche
  - Lille
  - Lyon
  - Nice
  - Paris
  - Pessac
  - Toulouse
  - Villejuif
- Germany (8):
  - Hanover, Niedersachesen
  - Bonn
  - Freiburg im Breisgau
  - Halle
  - Hamburg
  - Heidelberg
  - Leipzig
  - Mainz
- Hungary (4):
  - Debrecen
  - Gyula
  - Kaposvár
  - Pécs
- Israel (6):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Safed
  - Tel Aviv
- Italy (8):
  - Bergamo
  - Bologna
  - Florence
  - Milan
  - Palermo
  - Roma
  - Rozzano
  - San Giovanni Rotondo
- Netherlands (2):
  - Leiden
  - Maastricht
- Auckland, New Zealand
- Russia (2):
  - Moscow
  - Samara
- Spain (9):
  - A Coruña
  - Barcelona
  - Girona
  - Madrid
  - Málaga
  - Pontevedra
  - Santander
  - Seville
  - Valencia

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT01966419) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Safadi R, Rahimi RS, Thabut D, Bajaj JS, Ram Bhamidimarri K, Pyrsopoulos N, Potthoff A, Bukofzer S, Wang L, Jamil K, Devarakonda KR. Pharmacokinetics/pharmacodynamics of L-ornithine phenylacetate in overt hepatic encephalopathy and the effect of plasma ammonia concentration reduction on clinical outcomes. Clin Transl Sci. 2022 Jun;15(6):1449-1459. doi: 10.1111/cts.13257. Epub 2022 Mar 3. PMID 35238476
- [Derived] Wang X, Vilchez RA. Population Pharmacokinetic Analysis to Assist Dose Selection of the L-Ornithine Salt of Phenylacetic Acid. Clin Pharmacokinet. 2022 Apr;61(4):515-526. doi: 10.1007/s40262-021-01075-1. Epub 2021 Nov 17. PMID 34786649
- [Derived] Rahimi RS, Safadi R, Thabut D, Bhamidimarri KR, Pyrsopoulos N, Potthoff A, Bukofzer S, Bajaj JS. Efficacy and Safety of Ornithine Phenylacetate for Treating Overt Hepatic Encephalopathy in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Dec;19(12):2626-2635.e7. doi: 10.1016/j.cgh.2020.10.019. Epub 2020 Oct 16. PMID 33069881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 231 participants were enrolled (randomized) into the trial at multiple sites in the United States, Australia and Europe.
Groups:
- Placebo: Participants receive matching placebo up to 5 days via continuous IV infusion in addition to standard of care (SOC)
- Ornithine Phenylacetate: Participants receive ornithine phenylacetate for up to 5 days via continuous IV infusion in addition to SOC
Period: Overall Study
Arm/Group | Placebo | Ornithine Phenylacetate
Started | 115 | 116
Intent to Treat Population (ITT)T)115 | 115 | 116
Safety Analysis Set (SAS) | 112 | 114
Completed | 74 | 80
Not Completed | 41 | 36

BASELINE CHARACTERISTICS:
Population: Intent to treat population (ITT)
Groups:
- Ornithine Phenylacetate: Participants receive ornithine phenylacetate up to 5 days via continuous IV infusion in addition to SOC
- Total: Total of all reporting groups
Arm/Group | Placebo | Ornithine Phenylacetate | Total
Number analyzed (Participants) | 115 | 116 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.5) | 50 (9.8) | 59 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 81
  Male | 78 | 72 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 57 | 55 | 112
  Unknown or Not Reported | 51 | 50 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 5 | 13
  White | 54 | 59 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 51 | 50 | 101
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 4 | 5
  United States | 62 | 66 | 128
  Czechia | 4 | 1 | 5
  Russia | 7 | 5 | 12
  Spain | 3 | 10 | 13
  Austria | 2 | 5 | 7
  Netherlands | 1 | 0 | 1
  Belgium | 6 | 1 | 7
  Denmark | 2 | 0 | 2
  Italy | 0 | 2 | 2
  Israel | 11 | 11 | 22
  Australia | 1 | 0 | 1
  Bulgaria | 2 | 1 | 3
  France | 11 | 10 | 21
  Canada | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Each HE Stage
Description: To support the primary endpoint of confirmed clinical response, the investigator rated participants on a 4-point staging scale, where higher scores are worse.
  The stages are described as:
  Stage 0/1 = Participant has no tremor of the hand when the wrist is extended (asterixis) and no confusion, even about where they are (disorientation) Stage 2 = Participant has tremor of the hand when the wrist is extended (asterixis) and is confused, not knowing where they are (disorientation) Stage 3 = Participant is tired, falling asleep, answers questions but is confused, and doesn't know where they are (Stupor, arousable but falls asleep, responsive to verbal stimuli, Obvious confusion, Gross disorientation) Stage 4 = Participant is unconscious (in a coma)
Time Frame: Baseline to End of Study (through 3 hours post end-of-infusion)
Population: Intention to Treat Analysis Set (Note: all participants did not start at the same time)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ornithine Phenylacetate
Number analyzed (Participants) | 115 | 116
percentage of participants
  Baseline : Stage 4 | 11 | 6
  Baseline : Stage 3 | 30 | 40
  Baseline : Stage 2 | 71 | 68
  Baseline : Stage 0/1 | 0 | 0
  Baseline : Missing | 3 | 2
  Day 1, 7 am : Stage 4 | 0 | 0
  Day 1, 7 am : Stage 3 | 0 | 4
  Day 1, 7 am : Stage 2 | 2 | 3
  Day 1, 7 am : Stage 0/1 | 0 | 0
  Day 1, 7 am : Missing | 0 | 0
  Day 1, 5 pm : Stage 4 | 0 | 5
  Day 1, 5 pm : Stage 3 | 7 | 14
  Day 1, 5 pm : Stage 2 | 32 | 36
  Day 1, 5 pm : Stage 0/1 | 0 | 1
  Day 1, 5 pm : Missing | 0 | 0
  Day 2, 7 am : Stage 4 | 3 | 4
  Day 2, 7 am : Stage 3 | 21 | 15
  Day 2, 7 am : Stage 2 | 61 | 69
  Day 2, 7 am : Stage 0/1 | 10 | 10
  Day 2, 7 am : Missing | 0 | 0
  Day 2, 5 pm : Stage 4 | 3 | 4
  Day 2, 5 pm : Stage 3 | 14 | 9
  Day 2, 5 pm : Stage 2 | 57 | 61
  Day 2, 5 pm : Stage 0/1 | 16 | 16
  Day 2, 5 pm : Missing | 0 | 0
  Day 3, 7 am : Stage 4 | 3 | 2
  Day 3, 7 am : Stage 3 | 15 | 10
  Day 3, 7 am : Stage 2 | 50 | 55
  Day 3, 7 am : Stage 0/1 | 21 | 25
  Day 3, 7 am : Missing | 0 | 0
  Day 3, 5 pm : Stage 4 | 3 | 3
  Day 3, 5 pm : Stage 3 | 7 | 9
  Day 3, 5 pm : Stage 2 | 46 | 45
  Day 3, 5 pm : Stage 0/1 | 20 | 27
  Day 3, 5 pm : Missing | 0 | 0
  Day 4, 7 am : Stage 4 | 2 | 0
  Day 4, 7 am : Stage 3 | 5 | 9
  Day 4, 7 am : Stage 2 | 42 | 40
  Day 4, 7 am : Stage 0/1 | 28 | 30
  Day 4, 7 am : Missing | 0 | 0
  Day 4, 5 pm : Stage 4 | 2 | 0
  Day 4, 5 pm : Stage 3 | 5 | 7
  Day 4, 5 pm : Stage 2 | 42 | 34
  Day 4, 5 pm : Stage 0/1 | 28 | 28
  Day 4, 5 pm : Missing | 0 | 0
  Day 5, 7 am : Stage 4 | 0 | 0
  Day 5, 7 am : Stage 3 | 9 | 7
  Day 5, 7 am : Stage 2 | 29 | 28
  Day 5, 7 am : Stage 0/1 | 23 | 32
  Day 5, 7 am : Missing | 0 | 0
  Day 5, 5 pm : Stage 4 | 0 | 0
  Day 5, 5 pm : Stage 3 | 8 | 3
  Day 5, 5 pm : Stage 2 | 24 | 22
  Day 5, 5 pm : Stage 0/1 | 23 | 28
  Day 5, 5 pm : Missing | 0 | 0
  Day 6, 7 am : Stage 4 | 0 | 0
  Day 6, 7 am : Stage 3 | 10 | 3
  Day 6, 7 am : Stage 2 | 21 | 24
  Day 6, 7 am : Stage 0/1 | 23 | 27
  Day 6, 7 am : Missing | 0 | 0
  Day 6, 5 pm : Stage 4 | 0 | 0
  Day 6, 5 pm : Stage 3 | 3 | 3
  Day 6, 5 pm : Stage 2 | 5 | 7
  Day 6, 5 pm : Stage 0/1 | 6 | 5
  Day 6, 5 pm : Missing | 0 | 0
  End of Study : Stage 4 | 5 | 3
  End of Study : Stage 3 | 10 | 7
  End of Study : Stage 2 | 31 | 28
  End of Study : Stage 0/1 | 45 | 55
  End of Study : Missing | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 days
Description: Adverse events are reported in the safety population. All serious adverse events are reported. Non-serious treatment-emergent adverse events are reported at the 5% reporting threshold.
Arm/Group | Placebo | Ornithine Phenylacetate
All-Cause Mortality (participants affected / at risk) | 15/112 | 11/114
Serious Adverse Events (participants affected / at risk) | 34/112 | 29/114
Other Adverse Events (participants affected / at risk) | 31/112 | 30/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | Ornithine Phenylacetate (N=114)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 4 (4) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 2 (3) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 9 (9) | 9 (9)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 1 (1)
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | Ornithine Phenylacetate (N=114)
Anaemia (Blood and lymphatic system disorders) | 8 (11) | 13 (14)
Pyrexia (General disorders) | 7 (7) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10) | 9 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes